CLINICAL TRIAL: NCT03964714
Title: Monitoring Physical Activity in Acutely Hospitalized Elderly of 70 Years and Older
Acronym: MPA
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL65097.068.18
Record Dates: First submitted 2019-01-14; First posted 2019-05-28 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Physical Activity
Keywords: Acutely hospitalised; Elderly; Activity monitoring
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to create reference values regarding the amount of physical activity of acutely hospitalized elderly ≥70 years during hospitalization and aims to create a prediction model in order predict the probability of low amounts of physical activity of acutely hospitalized elderly ≥70 years during hospitalization.

DETAILED DESCRIPTION:
Rationale: Despite numerous studies supporting adverse outcomes associated with low physical activity (PA), there is insufficient insight in the amount of PA of acutely hospitalized Dutch elderly ≥ 70 years. PA can be objectively measured by accelerometers, but it is time consuming and expensive to provide every patient with an accelerometer. We need to be able to predict which elderly patients are likely to spend low amounts of physical activity during hospitalization. Because of the association between PA and functional decline it is expected that functional assessment tests like the Short Physical Performance Battery (SPPB) or Activity Measure for Post-Acute Care (AM-PAC) could be used as a screening tool to determine which patients will be at risk of low amounts of PA.

Objective: The primary objectives of this study are: 1) To assess the amount of PA of acutely hospitalized elderly ≥70 years during hospitalization and to create reference values regarding the amount of time patients are standing and walking per day and the number of breaks in sedentary time (BST) per day. 2) To be able to predict the probability of low amounts of physical activity during hospitalization for acutely hospitalized elderly ≥70 years.

Study design: This is a single center, observational, prospective cohort study.

Study population: 165 patients aged ≥70 years that are acutely hospitalized at the department of internal and geriatric medicine in the Maastricht University Medical Center (MUMC+).

Method: PA will be monitored with an accelerometer from inclusion (t0) until the day of intended discharge (t1). A functional assessment (SPPB and AM-PAC) will be performed at t0. Medical and demographic data will be obtained from the medical record and by patient report.

Main study parameters/endpoints: Mean number of minutes spent physically active (standing and walking) per day, dichotomized into a low and high amount of time spent physically active per day during hospitalization for the prediction model. Mean number of BST per day, dichotomized into a low and high number of BST per day during hospitalization for the prediction model.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Acutely hospitalized in MUMC+ at the department of Internal and Geriatric Medicine
* Sufficient understanding of the Dutch language
* Living at home before hospitalization
* Able to walk independently 2 weeks before admission, as scored on the Functional Ambulation Categories (FAC >3)

Exclusion Criteria:

* A life expectancy of less than three months as assessed by the attending physician
* Incapacitated subjects
* The inability to follow instructions due to cognitive problems or severe agitation
* A contraindication to wearing an accelerometer, fixated by a hypoallergenic plaster, on the upper leg (such as active bilateral upper leg infection, severe edema or bilateral transfemoral amputation)
* (Re)admittance to the intensive care unit
* Presence of contraindications to walking as assessed by the attending physician
* Previous participation to this study

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged ≥70 years that are acutely hospitalized in MUMC+ at the department of Internal and Geriatric Medicine.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2019-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Mean number of minutes spent physically active (standing and walking) per day | Measured continuously from the day of inclusion (Day 0) until the day the subject is medically ready to be discharged from the hospital.
  Defined as the total number of minutes standing and walking divided by the total number of valid measurement days in the period between inclusion and (intended) discharge. In order to create a prediction model, this will be dichotomized into a low and high amount of time spent physically active per day during hospitalization. As the estimated event rate of a high amount of time spent physically active per day during hospitalization is 50%, the cut-off value between a low and high amount of time spent physically active will be defined by dividing the cohort at the median.
Mean number of breaks in sedentary time (BST) per day | Measured continuously from the day of inclusion (Day 0) until the day the subject is medically ready to be discharged from the hospital.
  Defined as the total number of BST divided by the total number of valid measurement days in the period between inclusion and (intended) discharge. A BST is defined as any transition from being sedentary (lying or sitting) to being physically active (standing or walking).
  In order to create a prediction model, this will be dichotomized into a low and high number of breaks in sedentary time per day during hospitalization. As the estimated event rate of a high number of breaks in sedentary time per day during hospitalization is 50%, the cut-off value between a low and high number of breaks in sedentary time will be defined by dividing the cohort at the median.

SECONDARY OUTCOMES:
Short Physical Performance Battery scores (summary and component scores) | Measured on the day of inclusion (Day 0)
  Summary score on the scale: 0-12 points. Higher scores indicates better functioning. SPPB evaluates balance, gait, strength and endurance by examining an individual's ability to stand with feet together in side-by-side, semi-tandem and tandem positions, time to walk 4 meter and time to rise from a chair and return to the seated position five times. Component scores (0-4) for the three categories are measured as well.
Activity Measure for Post-Acute Care (AM-PAC) Inpatient Basic Mobility short form score | Measured on the day of inclusion (Day 0)
  The AM-PAC and provides a transparent measure of patients' capabilities in functional mobility during hospitalization. It measures the following daily activities: turning in bed, sitting down and standing up, moving from lying to sitting position, moving from a bed to a chair, walking and climbing stairs (6-24 points).
Age | Scored once on the day of inclusion (Day 0)
  Categories 70-79, 80-89, ≥90 years
Sex | Scored once on the day of inclusion (Day 0).
  Male / Female
Disability in activities of daily living (ADLs) two weeks prior to admission | Scored once the day of inclusion (Day 0).
  Number of disabilities on the Katz Index of Independence in Activities of Daily Living (Katz ADL). The Katz ADL measures the patient's ability to perform ADL independently. It is a dichotomous rating (dependant / independent) of six ADL functions, bathing, dressing, toileting, transferring, continence and feeding. It rates the level of independence or dependence in these tasks and is categorized by the amount of assistance needed to complete the task. The researcher will ask the patient how much assistance was needed to complete the tasks 2 weeks prior to admission.
The use of ambulation assistive devices prior to admission | Scored on the day of inclusion (Day 0).
  Yes/No. If yes, specify type of walking aid used prior to admission. The use of ambulation assistive device prior to admission is asked by the researcher.
Clinical diagnosis | On day of intended discharge from hospital, estimated up to 1 month. (Intended discharge is defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.)
  Clinical diagnosis as reported in the electronic medical record by the physician. The last reported clinical diagnoses by the physician before intended discharge will be extracted.
Physiotherapy consulted during hospitalization | On day of intended discharge from hospital, estimated up to 1 month. (Intended discharge is defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.)
  Did the patient receive one or more sessions of physiotherapy between inclusion and intended discharge? (Yes / No). All sessions will be reported by the physical therapist in the electronic medical record.

OTHER OUTCOMES:
History of falls in the past six months | Once, on the day of inclusion (Day 0)
  The number of falls in the last 6 months before hospital admission. Measured retrospectively by asking the patient the following question: Have you fallen once or more in the past six months? If yes, how many times? Question is asked by the researcher.
Medical comorbidities | On day of intended discharge from hospital, estimated up to 1 month. (Intended discharge is defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.)
  Charlson Comorbidity Index (CCI). Comorbidities are reported by the physician in the electronic medical record. All comorbidities present in the period between admission and intended discharge are extracted by the researcher and used to calculate the Charlson Comorbidity Index.
Length of stay | On day of intended discharge from hospital, estimated up to 1 month. (Intended discharge is defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.)
  Number of days from admission to the hospital to intended discharge (Defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.). Length of stay is retrieved from the electronic medical record.
Discharge location | On day of intended discharge from hospital, estimated up to 1 month. (Intended discharge is defined as the day the patient is medically ready for discharge and is either discharged or staying for non-medical reasons.)
  Home, geriatric rehabilitation center, nursing home, other. As reported in the electronic medical record by the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine F Lenssen, Prof., PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown CJ, Roth DL, Allman RM. Validation of use of wireless monitors to measure levels of mobility during hospitalization. J Rehabil Res Dev. 2008;45(4):551-8. doi: 10.1682/jrrd.2007.06.0086. PMID 18712640
- [Result] Evensen S, Sletvold O, Lydersen S, Taraldsen K. Physical activity among hospitalized older adults - an observational study. BMC Geriatr. 2017 May 16;17(1):110. doi: 10.1186/s12877-017-0499-z. PMID 28511639
- [Result] Fisher SR, Goodwin JS, Protas EJ, Kuo YF, Graham JE, Ottenbacher KJ, Ostir GV. Ambulatory activity of older adults hospitalized with acute medical illness. J Am Geriatr Soc. 2011 Jan;59(1):91-5. doi: 10.1111/j.1532-5415.2010.03202.x. Epub 2010 Dec 16. PMID 21158744
- [Result] Ostir GV, Berges IM, Kuo YF, Goodwin JS, Fisher SR, Guralnik JM. Mobility activity and its value as a prognostic indicator of survival in hospitalized older adults. J Am Geriatr Soc. 2013 Apr;61(4):551-7. doi: 10.1111/jgs.12170. Epub 2013 Mar 25. PMID 23527951
- [Result] Pedersen MM, Bodilsen AC, Petersen J, Beyer N, Andersen O, Lawson-Smith L, Kehlet H, Bandholm T. Twenty-four-hour mobility during acute hospitalization in older medical patients. J Gerontol A Biol Sci Med Sci. 2013 Mar;68(3):331-7. doi: 10.1093/gerona/gls165. Epub 2012 Sep 12. PMID 22972940